CLINICAL TRIAL: NCT06878859
Title: AMP-C: A Digital Therapeutic for Reward Dysfunction in Co-Occurring Depression and Cannabis Use
Brief Title: Preliminary Efficacy Trial of a Digital Intervention for Depression and Cannabis Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Amanda C. Collins, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025p000583; 1K23DA062034 (NIH)
Record Dates: First submitted 2025-03-06; First posted 2025-03-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; Cannabis Use Disorder; Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amplification of Positivity - Cannabis Use (AMP-C) (Experimental)
  Interventions: Behavioral: Amplification of Positivity - Cannabis Use (AMP-C)
- Symptom Tracking (No Intervention)

INTERVENTIONS:
Behavioral: Amplification of Positivity - Cannabis Use (AMP-C) — AMP-C is a smartphone-based digital intervention that includes activities that focus on positivity (e.g., noticing and capitalizing on positive events) to increase positive emotions, thoughts, and behaviors. The role and impact of CU on the maintenance of depression and reward dysfunction (and vice versa), is intertwined throughout the intervention.
  Arms: Amplification of Positivity - Cannabis Use (AMP-C)

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability, and preliminary efficacy of a digital intervention for co-occurring cannabis use and depression. Participants will be randomized to complete Amplification of Positivity - Cannabis Use (AMP-C) or symptom tracking. The main outcomes will include changes in depressive symptoms and cannabis use, as well as usability ratings.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Resides in the United States
* Able to read and understand English and willing to provide informed consent/comply with the study protocol
* Moderate depressive symptom severity, as indicated by the Patient Health Questionnaire-9 (PHQ-9)
* Problematic cannabis use, as indicated by the Cannabis Use Disorder Identification Test - Revised (CUDIT-R)
* Current elevated anhedonia, as indicated by the PHQ-9
* Interest in receiving treatment for their cannabis use and depression
* Meet criteria for current MDD and CUD per the DSM-5

Exclusion Criteria:

* History of a psychotic disorder or bipolar disorder type I/II
* Active suicidal ideation or intent based on the Columbia-Suicide Severity Rating Scale
* Current psychotherapy engagement
* Changes in psychotropic medication within six weeks of the start of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms (Patient Health Questionnaire-9; PHQ-9) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: Intervention Midpoint (4 weeks into intervention), 1-, 3-, 6-, and 12-months after completing intervention
  Depressive symptoms will be measured with the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a widely-used 9-item self-report measure that assesses depressive symptom severity over the previous two weeks. Scores on the PHQ-9 range from 0-27, with greater scores indicating greater depression severity.
Change in Cannabis Use Frequency (Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory; DFAQ-CU) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: Intervention Midpoint (4 weeks into intervention), 1-, 3-, 6-, and 12-months after completing intervention
  Cannabis use use will be measured with the Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory (DFAQ-CU). The DFAQ-CU is a 24-item self-report measure that assesses frequency, age of onset, and quantity of cannabis use. There are six factors: daily sessions, frequency, age of onset, marijuana quantity, concentrate quantity, and edible quantity. The six factors, except age of onset, are independently scored, and higher scores indicate greater cannabis use. Our primary outcome will assess changes in frequency.
Usability (System Usability Scale; SUS) | Post-Intervention (approximately one week after completing intervention)
  The System Usability Scale (SUS) is a 10-item self-report measure commonly used to assess the degree to which participants endorse ease of use following task-based operation of computer systems (i.e., perceived usability). Total scores on the SUS range from 0 to 100, with greater scores indicating greater usability. An average score of 68 or greater on the SUS in our AMP-C group will indicate acceptable usability.

SECONDARY OUTCOMES:
Feasibility (Engagement) | Post-Intervention (approximately one week after completing intervention)
  Feasibility will be measured through the number of modules completed for the AMP-C group.
Intervention Feasibility (App Usage) | Post-Intervention (approximately one week after completing intervention)
  Feasibility will be measured through app usage time (hours).
Change in Daily Depressive Symptoms (Mobile Patient Health Questionnaire-9; MPHQ-9) | Daily for 8 weeks during intervention
  Daily depressive symptoms will be measured with the Mobile Patient Health Questionnaire-9 (MPHQ-9). The MPHQ-9 is a modified version of the paper PHQ-9, which has been used in intensive sampling studies. Participants answer questions regarding their experience with the nine symptoms of MDD over the past 24 hours on a sliding scale. Total scores range from 0-900, with greater scores representing greater depression severity.
Changes in Daily Cannabis Use | Daily for 8 weeks during intervention
  Daily cannabis use will be measured with a series of questions related to cannabis use consumption. These questions will capture frequency, quantity, product types, potencies, and administration methods of cannabis over the past 24 hours.
Change in Positive Affect (Positive and Negative Affect Schedule-Positive Affect; PANAS-PA) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: Intervention Midpoint (4 weeks into intervention), 1-, 3-, 6-, and 12-months after completing intervention
  The Positive and Negative Affect Schedule Scale-Positive Affect (PANAS-PA) is a 10-item self-report measure that assesses positive affect over the past week. Total scores range from 10-50, with greater scores representing greater positive affect.
Change in Anticipatory and Consummatory Anhedonia (Temporal Experience of Pleasure Scale; TEPS) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  Anticipatory and consummatory anhedonia will be measured with the Temporal Experience of Pleasure Scale (TEPS). The TEPS is a 18-item self-report measure that assesses reward anticipation (e.g., motivation) and responsiveness (e.g., pleasure). There are two subscales in the TEPS: anticipatory anhedonia and consummatory anhedonia. Scores on the anticipatory subscale range from 10 to 60, and scores on the consummatory subscale range from 8 to 48. Higher scores indicate greater pleasure.
Change in Negative Affect (Positive and Negative Affect Schedule-Negative Affect; PANAS-NA) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  The Positive and Negative Affect Schedule Scale-Negative Affect (PANAS-NA) is a 10-item self-report measure that assesses negative affect over the past week. Total scores range from 10-50, with greater scores representing greater negative affect.
Changes in passive sensing behaviors | Continuously for 8 weeks during intervention
  Passive sensing behaviors will be continuously collected without requiring participant input and will be related to psychomotor agitation (measured through high-frequency oscillations from daytime accelerometer activity), sleep disturbances (measured through nighttime accelerometer activity, GPS location, and screen unlocks), behavioral activation (measured through GPS mobility), social contact (measured through timestamps and duration of calls, texts, and in-person conversations (i.e., not the actual content of calls, messages, or conversations), exposure to natural light (measured through light sensors), and screen time (measured through app usage). Changes in behaviors (e.g., increased GPS mobillity) will indicate greater behavioral activation during the course of the intervention for the AMP-C group.

OTHER OUTCOMES:
Change in Alcohol Use (Drinking Motives Questionnaire-Revised; DMQR) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  Reasons for drinking alcohol will be measured with the Drinking Motives Questionnaire-Revised (DMQR). The DMQR is a 20-item self-report measure that assesses common reasons for why people might drink alcohol. There are four subscales: Social, Coping, Enhancement, and Conformity. Subscale scores range from 1-25, with greater scores representing greater endorsement of specific reasons for drinking alcohol.
Change in Substance Use (Timeline Followback; TLFB) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  Broader substance use will be measured with the Timeline Followback (TLFB). The TLFB is a self-report measure that assesses substance use and related behaviors over the past 30 days. Participants will be asked to identify the number of days over the 30 days in which they have consumed alcohol, tobacco/nicotine, opioids, stimulants, hallucinogens, sedatives/depressives, inhalants, and other illicit or prescription drugs. Total scores are not calculated, but the outcomes of interest include number of days per substance, with greater scores indicating a higher number of days of substance use in the past 30 days.
Change in Anxiety Symptoms (Generalized Anxiety Disorder-7; GAD-7) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  Anxiety symptoms will be measured with the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 is a 7-item self-report measure that assesses anxiety symptom severity over the previous two weeks. Total scores range from 0-21, with higher scores representing higher anxiety severity.
Change in Fear of Happiness (Fear of Happiness Scale; FHS) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  The Fear of Happiness Scale (FHS) is a 9-item self-report measure that assesses fear and apprehension of positivity due to its association with negative outcomes. Total scores range from 0-36, with greater scores representing greater fear of happiness.
Change in Dampening (Responses to Positive Affect Scale) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  Dampening will be measured with the Responses to Positive Affect Scale (RPA; RPA) is a widely-used 17-item self-report measure that assesses dampening and amplifying of positive emotions. Scores on dampening subscale range from 8-32, with greater scores indicating greater dampening.
Change in Well-Being (Warwick-Edinburgh Mental Wellbeing Scale; WEMWBS) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) is a 14-item self-report measure developed to capture positive aspects of mental health in the general population. Participants indicate how often over the past two weeks they have experienced each statement on a five-point Likert scale ranging from 1 ("None of the time") to 5 ("All of the time"). Total scores range from 14 to 70, and greater scores reflect greater overall mental well-being.
Change in Social Connectedness (Social Connectedness Scale - Revised; SCS-R) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  The Social Connectedness Scale - Revised (SCS-R) is a 20-item self-report measure that assesses individuals' sense of interpersonal closeness and belongingness with others. It captures the extent to which people feel emotionally connected to, understood by, and integrated within their social world. The SCS-R will be used to evaluate participants' perceived social connectedness and sense of belonging as an indicator of social and emotional well-being. Scores range from 20-120, with greater scores indicating greater social connectedness.
Change in Reward Devaluation (Valence Selection Task; VST) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  The Valence Selection Task (VST) is a behavioral paradigm designed to assess cognitive-emotional biases in the processing of affective information, based on principles from Reward Devaluation Theory (RDT). The task involves presenting participants with incomplete reading prompts and requiring them to choose between three plausible sentence endings that differ in emotional valence, namely positive, negative, or neutral. This setup models a naturalistic decision-making scenario, akin to everyday reading or interpretation of emotional content. Outcome indices include propotion of positive, negative, or neutral choices selected, with lower proportion of selecting positive responses indicating greater reward devaluation.
Change in Positive Self-Schemas (Self-Referent Encoding Task; SRET) | Baseline, Primary Endpoint: Post-Intervention (approximately one week after completing intervention), Secondary Endpoints: 1-, 3-, 6-, and 12-months after completing intervention
  The Self-Referent Encoding Task (SRET) is a cognitive measure that assesses self-schemas and biases in processing emotional information. Participants view positive and negative adjectives and indicate whether each describes them ("Describes me?"), followed by a recall phase. The SRET evaluates endorsement, recall, and reaction time for self-referential words. Consistent with Reward Devaluation Theory, depressed individuals typically endorse and recall fewer positive and more negative self-descriptive words. The SRET will be used to assess self-referential processing and devaluation of positivity as indicators of cognitive-emotional functioning. Primary outcomes will include number of reponses of (1) "yes" and (2) "no" to self-referential positive words, with greater number of words for the former (1) indicating positive self-schemas and greater number of words for the latter (2) indicating devaluative self-schemas.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No